CLINICAL TRIAL: NCT03724682
Title: A Performance Analysis of the Peritoneal Ultrafiltration (PUF) Achieved With the Carry Life® UF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triomed AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tmed-007 (Malmö)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-10

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Baseline study session with standard PD therapy. Three study sessions with the Carry Life UF device at three different glucose dosages, starting with the lowest dose of 11g/h, increasing to 14g/h and finally 20g/h.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm in which everyone enrolled in a trial receives treatment with Carry Life UF device,
  Interventions: Device: Carry Life UF device

INTERVENTIONS:
Device: Carry Life UF device — Treatment with the Carry Life UF device compared to standard PD therapy

SUMMARY:
The Carry Life UF device performs peritoneal ultrafiltration by adding a concentrated glucose to peritoneal dialysis fluid which has been instilled into the abdomen prior to the connection of the device. Maintaining the glucose concentration in the intraperitoneal fluid results in an increased fluid removal (ultrafiltration).

The clinical investigation will evaluate the ultrafiltration achieved with the Carry Life UF device compared to standard peritoneal dialysis (PD) therapy

DETAILED DESCRIPTION:
A study of the peritoneal ultrafiltration achieved with Carry Life® UF compared to standard PD therapy, performed in 12 stable PD patients. The study consists of one baseline study session with Icodextrin overnight and one four-hour, 2.27% glucose exchange and three Carry Life® UF treatments with different glucose doses. All treatments are preceded by an Icodextrin dwell overnight.

Visit 1: The patient will be screened for study eligibility and a signed informed consent obtained before any of the study activities commence. Once included in the study the patient will be asked to document their ultrafiltration volumes for the week prior to the baseline study session (PD bags to be weighed before and after).

Visit 2: Baseline study session with standard PD therapy. The evening before visit 2 the patient will use Icodextrin 2000 ml overnight which is drained at the clinic before the start of the second PD exchange.

* A four-hour dwell with 2.27%, 2000 ml PD fluid will be performed at the clinic.
* During the study sessions the fluid intake and output will be measured.
* A 24 h urine collection for urea and creatinine clearance started the day before the baseline study session will be completed at the baseline study session.

Visit 3, 4 and 5: Carry Life® UF study sessions The evening before the visits the patient will use Icodextrin 2000 ml overnight which is drained at the clinic the next day before the start of the Carry Life® UF study session.

* The Carry Life UF study session starts with filling the peritoneal cavity with 1500 ml of a standard glucose-based PD solution of 1.36%.
* The Carry Life® UF is then connected to the PD catheter and the 5-hour treatment starts. The glucose dose for visit 3 is 11 g/h, visit 4, 14 g/h and visit 5, 20 g/h.
* During the treatment, IP fluid will be drained hourly and as required.
* During the study sessions the fluid intake and output will be measured.
* During and after each study session the patient's tolerability of the treatment will be evaluated by monitoring vital signs (blood pressure and heart rate hourly).
* Evaluation of the patient's experience of the Carry Life® UF treatment is documented in the CRF, regarding the sensation of the flow in and out of the abdomen and a short questionnaire between visit 4 and 5, regarding the usability and experience of the device.

Follow-up: Follow-up will be performed after the completion of the Carry Life® UF study sessions. The follow-up can either be performed at the clinic or by telephone which is at the discretion of the investigator and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Male or female
* On stable PD including Icodextrin, treated at the clinic for at least 3 months
* No clinical signs of dehydration.
* Obtained written consent to participate in the study

Exclusion Criteria:

* Significant illness or active infection (evaluated by clinical examination) in the past 4 weeks
* Episodes of peritonitis during the past 2 months
* Active malignant disease
* Diabetes type 1
* Abdominal hernias
* HIV and/or hepatitis positive within the last 3 months
* Known pregnancy or breastfeeding and pregnancy test for women of child bearing age.
* Conditions deemed by investigator as inappropriate for participation
* Participation in clinical trials, interfering with the present study, one month prior to inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Ultrafiltration volume | During a five hour study session
  The ultrafiltration volumes achieved during the study sessions

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrine Johansson, Principal Investigator — Renal Unit, Skånes Universitetssjukhus, Malmö
Locations (3):
- Sweden (3):
  - Skånes Universitetssjukhus, Malmö, Malmo, Skåne County
  - Skånes Universitetssjukhus, Lund, Lund
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No
The results of the investigation will be submitted for publication, and publications and presentations will be based upon the clinical investigation report.

REFERENCES:
- [Derived] Heimburger O, Hegbrant J, Martus G, Wilkie M, De Leon C, Carlsson O, Johansson AC. Effects of Steady Glucose Concentration Peritoneal Dialysis on Ultrafiltration Volume and Sodium Removal: A Pilot Crossover Trial. Clin J Am Soc Nephrol. 2024 Feb 1;19(2):224-232. doi: 10.2215/CJN.0000000000000342. Epub 2023 Oct 30. PMID 37902732